CLINICAL TRIAL: NCT05072704
Title: Opioid Free Anesthesia in Total Hip Arthroplasty. A Randomized, Controlled and Triple-blind Clinical Trial
Brief Title: Opioid Free Anesthesia in Total Hip Arthroplasty
Acronym: OFATHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/04
Record Dates: First submitted 2021-09-17; First posted 2021-10-11 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: Hip arthroplasty; Opioid free anesthesia; Dexmedetomidine; Postoperative analgesia
MeSH Terms: interventions — Sufentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Sufentanil IV injection
  Interventions: Drug: Sufentanil
- OFA group (Experimental): Dexmedetomidine IV infusion
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Sufentanil — Pre-operative injection of sufentanil 10µg in 2ml of normal saline on induction of anesthesia + per-operative injection of sufentanil 5µg in 1ml of normal saline during the surgery if needed.
  Arms: Control group
Drug: Dexmedetomidine — Pre-operative infusion of dexmedetomidine 1µg/kg in 100ml of normal saline before surgery + per-operative infusion of dexmedetomidine 0.4 µg/kg in 100ml of normal saline during the surgery if needed.
  Arms: OFA group

SUMMARY:
Total hip arthroplasty (THA) is one of the most common orthopedic surgical procedure and is associated with severe pain in the immediate postoperative period, thus limiting early recovery.

Postoperative pain management in THA requires multimodal analgesia, combining drugs and injection of a local anesthetic (LA). But, the best anesthesia strategy to provide optimal postoperative analgesia in THA remains controversial. Opioid free anesthesia could limit the episodes of hyperalgesia as well as tolerance and addiction to opioids.

The hypothesis of this study is that an opioid free anesthesia using dexmedetomidine could improve analgesia after THA.

The main objective of this monocenter, prospective, randomized, triple-blind, controlled trial is to assess the interest of opioid free anesthesia using dexmedetomidine on morphine consumption after THA.

DETAILED DESCRIPTION:
In the pre-anaesthesia room, after the implementation of classical monitoring and a peripheral venous catheter, all patients will receive an antibioprophylaxis according to SFAR (French Society of Anesthesia & Intensive Care Medecine) recommendations and injection of 10 mg of IV dexamethasone.

The patients will be then randomized in 2 groups:

Control group:

* Pre-operative normal saline infusion 100 ml over 30 minutes
* Injection of sufentanil 10 µg in normal saline 2 ml on induction of anesthesia

If needed after incision :

* Per-operative normal saline infusion 100 ml
* Per-operative injection of sufentanil 5 µg in normal saline 1 ml

OFA group (experimental group):

* Pre-operative dexmedetomidine infusion 1 µg/kg in normal saline 100 ml over 30 minutes
* Injection of normal saline 2 ml on induction of anesthesia

If needed after incision :

* Per-operative dexmedetomidine infusion 0.4 µg/kg in normal saline 100 ml
* Per-operative injection of normal saline 1 ml

In the operating room, general anesthesia will be induced by intravenous ketamine (0.4 mg/kg) + propofol (3 mg/kg) +/- cisatracurium (0.1 mg/kg) for the introduction of laryngeal mask airway. Anesthesia will be maintained with propofol.

Postoperative analgesia protocol :

* Multimodal analgesia will be instituted during surgery by the administration of paracetamol (1 g), nefopam (20 mg) and ketoprofen (100 mg) and the infiltration of the surgical wound with 100 ml of ropivacaine 0.2%.
* In post-anesthesia care unit (PACU): oxycodone titration if NRS (pain score) >3 according to the centre's usual care.
* In ward and at home: systematic per os analgesia with paracetamol (1 g, 4 times a day) and ibuprofen (400 mg, 3 times a day); oxycodone (10 mg, lockout interval: 4 h) if NRS (pain score) >3.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Undergoing outpatient primary total hip arthroplasty under general anesthesia with laryngeal mask,
* Consent for participation,
* Affiliation to a social security system

Exclusion Criteria:

* Heart rate < 60 bpm
* Chronic pain syndrome requiring preoperative morphine use (class 3)
* Contraindication for: paracetamol, ketoprofen, nefopam, oxycodone, propofol, ketamine, cisatracurium, sufentanyl, ropivacaine.
* Contraindication for dexmedetomidine: hypersensitivity to the active substance or to any of the excipients, advanced cardiac block (grade 2 or 3) unless paced ; uncontrolled hypotension ; acute cerebrovascular conditions
* Contraindication to laryngeal mask : old insulin-dependent diabetes, gastro-oesophageal reflux, morbid obesity (defined by BMI > 35)
* Pregnant or breastfeeding women
* Women of child bearing potential without contraception (any contraceptive method used regularly and appropriately with a low failure rate: <1% per year),
* A mental or linguistic inability to understand the study,
* Patient under protection of the adults (guardianship, curators or safeguard of justice),
* Patient included or planning to be included in another clinical trial relating to medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia, defined by the oxycodone consumption in the first 24 hours post-surgery | 24 hours
  Postoperative cumulated dose of oxycodone in oral morphine equivalent (mg)

SECONDARY OUTCOMES:
Analgesia in post-anesthesia care unit (PACU) | 6 hours
  Total amount of oxycodone (mg) administered in PACU
Postoperative pain at rest | 24 hours
  Postoperative pain at rest (numeric rating scale ranging from 0 to 10: 0= no pain; 10= worst imaginable pain)
Postoperative pain at walk | 24 hours
  Postoperative pain at mobilization (numeric rating scale ranging from 0 to 10: 0= no pain; 10= worst imaginable pain)
Side effects associated with opioids | 24 hours
  Complications due to oxycodone (postoperative nausea and vomiting, drowsiness, acute urinary retention, pruritus, disorientation)
Side effects associated with dexmedetomidine | 24 hours
  Complications due to dexmedetomidine (bradycardia defined by HR<50 bpm or requiring the use of atropine; hypotension defined by SBP<90 mmHg or requiring the use of vasoconstrictors; hypertension defined by SBP>160 mmHg).
Outpatient care failure | 24 hours
  Unplanned hospitalizations
Length of stay in post-anesthesia care unit (PACU) | 6 hours
  Duration of PACU stay (min)
Time to recover the ability to walk | 12 hours
  Duration for recovery the ability to walk (min)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Médipôle Garonne, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No